CLINICAL TRIAL: NCT06540300
Title: Effects of Repetitive Transcrannial Magnetic Stimulation on Non-Suicidal Self-Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, Associate chief physician, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-KY035-01
Record Dates: First submitted 2024-07-10; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: NSSI

STUDY DESIGN:
Intervention Model Description: This study used a randomized, double-blind study method that controlled true and false stimuli. Except for the study leader, neither the actual operators nor the patients themselves knew whether they were receiving real or fake stimuli.
  A two factor mixed trial design was adopted, with a detection time of 2 (pre stimulus vs post stimulus) x 2 (stimulus type: right IPL vs pseudo stimulus). The stimulus type was an inter subject factor, and the detection time was an intra subject factor.
  The enrolled NSSI patients were randomly divided into a study group (right IPL group) and a control group (pseudo stimulus group) using a random number table method. Collect general demographic scales, symptom scales, and magnetic resonance imaging data before treatment, and conduct symptom scale retesting and magnetic resonance imaging data collection 2 weeks after treatment.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effects of rTMS on NSSI (Experimental): Exploring the effectiveness of rTMS intervention in NSSI patients using the Ottawa Self Injury Scale and other scales as research subjects
  Interventions: Other: rTMS stimulation of right IPL
- rs-fMRI-functional connectivity (Experimental): Based on rs fMRI technology, imaging methods were used to analyze the brain images of patients and explore the changes in functional connectivity of brain regions before and after intervention in two groups of subjects.
  Interventions: Other: rTMS stimulation of right IPL

INTERVENTIONS:
Other: rTMS stimulation of right IPL — The stimulation site is the right IPL (EEG International 10-20 system, electrode CP4/CP6), with a stimulation frequency of 1-Hz and intensity of 100% RMT. There are 50 pulses each time, 20 seconds each cycle, 5 seconds each, with an interval of 15 seconds, for a total of 60 cycles, a total duration of 20 minutes, and a total of 3000 pulses. Perform treatment once a day, rest for 2 days after 5 consecutive days of treatment, for a total of 2 weeks, and receive 10 treatments.

SUMMARY:
Non-suicidal self-injury (NSSI) refers to a series of direct and consequently repeated injuries to one's body without suicidal intent. At present, it has become an important issue of mental disorders. This article focuses on the formation mechanism of NSSI and the intervention effect of rTMS on NSSI patients. At the same time, NSSI patients are collected, a treatment plan is designed to complete a two-week treatment, and the results are analyzed. The aim is to provide theoretical basis for the clinical diagnosis and treatment of NSSI, and also to provide reference for the clinical diagnosis and treatment of NSSI patients.

DETAILED DESCRIPTION:
Research Objective Non suicidal self injury (NSSI) behavior is a common behavioral issue in psychiatric and psychiatric clinics. Studies have shown that NSSI is on the rise in China and has become an important mental health issue. Non suicidal self injury and suicide have similar clinical manifestations. Therefore, this study will intervene in the treatment of NSSI patients, understand the occurrence of NSSI in psychiatric outpatient and inpatient wards, and observe the efficacy of repeated transcranial magnetic stimulation intervention in NSSI patients, in order to explore the current occurrence status and biopsychological etiology of NSSI in psychiatric clinical practice.

Research Process If you agree to participate in this study, please read and sign this informed consent form before participating in any of the following procedures.

Research location: All research processes and evaluation interviews were conducted at the Affiliated Brain Hospital of Nanjing Medical University.

Study participants: Participants clinically diagnosed with non suicidal self injury participated in this study, aged 10-60 years, regardless of gender. All participants entered the study after signing the informed consent form.

Research Procedures This study first clarifies your diagnosis by conducting interviews to understand your physical health status, course of illness, family history, previous medical treatment, and examination results. We will assign a number to each participant, establish a medical record, and then perform corresponding psychological assessments, magnetic resonance imaging examinations, and repeat transcranial magnetic stimulation therapy for two weeks (a total of 10 times).

Possible Benefits All clinical scale evaluations, imaging examinations, and repeated transcranial magnetic stimulation interventions related to the study are free of charge. Your research doctors and evaluators will conduct timely clinical observations of changes in your condition, and provide you with systematic research follow-up and evaluation. These evaluations will help make reasonable judgments about your disease status and treatment effectiveness, and thus guide treatment decisions more scientifically. In addition, free treatment with repeated transcranial magnetic stimulation is also beneficial for the improvement of your condition. The research team will coordinate with relevant staff in the hospital and department where you are seeking medical treatment to provide convenience in basic clinical services such as doctor appointments, registration, and waiting, in order to save your visit time.

Privacy and Confidentiality Issues If you decide to participate in this study, your participation in the experiment and your personal information during the experiment will be kept confidential. Responsible research doctors and other researchers will use your medical information for research, but will not disclose your personal information. If you are harmed by participating in this study, you can receive free treatment and/or corresponding compensation.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the NSSI diagnostic criteria recommended in DSM-5;
2. The Chinese version of the Brief International Neuropsychiatric Interview (MINI) screen for diagnostic compliance;
3. Age :10-55 years old;
4. Right hand;
5. The paitent voluntarily participate and sign the informed consent form for this study (signed by participants under the age of 18 and their families);
6. Able to understand written language and cooperate with questionnaire surveys.

Exclusion Criteria:

1. History of severe substance abuse;
2. The patient has other serious mental disorders, neurological disorders, or physical illnesses; 3、Previously experienced epileptic seizures;

4、Pregnant or lactating women; 5、Contraindications to magnetic resonance imaging and transcranial magnetic stimulation; 6、Unable or refused to provide written informed consent.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Ottawa Self-injury Inventory | 2 weeks
  OSI was evaluated by professionally trained doctors (non experimental intervention) at baseline and two weeks after treatment to assess the effectiveness of the treatment. Comparing the differences in self harm thoughts and behaviors between the baseline period and the intervention group and the control group, p<0.05 indicates a significant difference.
Magnetic resonance imaging | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided